CLINICAL TRIAL: NCT00331890
Title: Citicoline in the Treatment of Acute Ischemic Stroke. An International Randomized Multicenter Placebo-controlled Study
Brief Title: ICTUS Study: International Citicoline Trial on Acute Stroke
Acronym: ICTUS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: With 2078 patients, a statistical stopping boundary has now been crossed
Sponsor: Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GF-ICTUS-04
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Acute Stroke; Cerebral Infarction
Keywords: Neuroprotection; Acute ischemic stroke; Cerebral infarction
MeSH Terms: conditions — Stroke; Cerebral Infarction; Ischemic Stroke | interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): Receives active drug
  Interventions: Drug: Citicoline
- Placebo (Placebo Comparator): Receives a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citicoline — 1g/12h iv during 3 days and then orally until complete 6 weeks of treatment
  Other Names: CDP-choline
  Arms: Active
Drug: Placebo — As active drug
  Arms: Placebo

SUMMARY:
Citicoline is a safe drug approved in some countries for the treatment of acute ischemic stroke. The drug has shown some evidence of efficacy in a pooled analysis, based on four clinical trials done in USA with oral citicoline.The purpose of the study is confirm the results obtained in the pooled analysis, that is, evidence of efficacy in the treatment of acute ischemic stroke

DETAILED DESCRIPTION:
The stroke or brain attack is one of the main health problems in developed countries. It is the third cause for death and the main cause of disability in adults. Cerebral infarction makes up 80 % of all the types of strokes.

After a stroke, different evolutions and outcomes can be observed, and there are several factors that may influence the outcome, such as age, cognitive impairment, and psycho-social factors. The most important prognostic factors for acute ischemic stroke are the volume of the cerebral infarction and the severity of the baseline neurological deficit.

In recent years, stroke has been considered a real medical emergency, and for this reason several clinical trials have been conducted to find effective therapies. Among pharmacological therapies, there are two possible ways to treat ischemic strokes: treatments directed to recanalize the occluded artery, such as thrombolysis, and the neuroprotective drugs.

None of the neuroprotective drugs have attained the international approval for this indication. Among the reasons for the failures obtained with the different drugs tested, we must highlight the problems derived from the toxicity of the drugs and from the evaluation criteria, as well as the therapeutic window used.

To evaluate a drug in the treatment of acute ischemic stroke, one must be very careful when defining the schedule of the clinical trial, and which variable or variables may be considered as primary endpoints. Several endpoints have been used in the different clinical trials developed, although the most used are those referring to the functional status and the degree of disability of the patients, normally set at 3 months after the stroke.

After the onset of an ischemic stroke in the brain, there is a cascade of events that are responsible for neuronal disruption, neuronal membrane breakdown and/or neuronal apoptosis, specifically in the penumbra area. Therapies acting by blocking the ischemic cascade, at least partially, and/or stabilizing neuronal membranes are believed to be beneficial protecting the brain from the progressive effects of ischemia. Among the neuroprotective drugs, there is a new class of drugs, of which the main representative is citicoline. Citicoline monosodium is an exogenous form of CDP-Choline, which is essential for the biosynthesis of membrane phospholipids. The mechanisms of action of citicoline include the stimulation of the biosynthesis of phospholipids of the neuronal membrane, the inhibition of the activity of some phospholipases, the restoration of some enzymatic activities bound to neuronal membranes, and the elevation of brain levels of some catecholamines.

The previous clinical trials performed with citicoline were no conclusive, with some positive results. In all these studies, citicoline was found to have a similar safety profile as compared with placebo.

The variety of outcomes and results of the different trials made it difficult to arrive at a consensus on the efficacy of the drug. That is the reason why a Pooling Data Analysis using updated individual patient data was done, with the main objective to determine the effects of citicoline on the improvement, functional and neurological, of patients with acute ischemic stroke treated with different doses of citicoline for 6 weeks and with a follow-up period of 6 weeks. The results obtained in this Pooling Data Analysis showed that the odds ratio of achieving a complete recovery was 33 % higher in citicoline-treated patients than in placebo-treated patients, with the best response obtained with the dose of 2000 mg/d/6 weeks.

The primary objective of this study is to determine the effects on recovery at 3 months of oral citicoline 2000 mg/d/6 weeks, after 6 weeks of treatment and 6 weeks of follow-up, in patients with moderate-to-severe acute ischemic strokes (baseline NIHSS equal or higher than 8) in comparison with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, >18 years old
* Patients must be treated within 24 hours of their initial stroke symptoms onset.
* Patients with a measurable focal neurological deficit lasting for a minimum of 60 minutes.
* Patients must have a CT scan and/or conventional MRI compatible with the clinical diagnosis of acute ischemic stroke prior to being randomized.
* Patients must have an acute ischemic stroke referable to the middle cerebral artery territory
* At inclusion, NIHSS score > 7, with at least 2 of these points from sections 5 & 6 (motor)
* Immediately (i.e. minutes) pre-stroke, MRS < 2
* Women of childbearing potential must have a negative pregnancy test prior to enrolment
* Signed informed consent

Exclusion Criteria:

* Patients in coma: patients having a score of 2 or higher in the items regarding the level of consciousness in the NIHSS (1a)
* CT or conventional MRI evidence of brain tumor, cerebral edema with a clinically significant mass midline shift with compression of the ventricles, brainstem or cerebellar infarction, subarachnoid and/or intracerebral and/or intraventricular hemorrhage
* History of ventricular dysrhythmias, acute myocardial infarction within 72 hours prior to enrolment, unstable angina, decompensated congestive heart failure or any other acute, severe, uncontrollable or sustained cardiovascular condition that, in the Investigator's opinion, may interfere with effective participation in the study
* Previous disorders that may confound the interpretation of the neurological scales
* Drug addiction-related disorders
* Pre existing dementia, when dementia implies a disability, measured as an score of 2 or higher in the previous MRS
* Pre existing medical condition that, in the Investigator's opinion, may interfere with the patient's suitability and participation in the study
* Patients participating in another clinical trial or receiving a non-approved drug (clinical investigational drug) less than 30 days prior to screening
* Patients under current treatment with citicoline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2298 (Actual)
Dates: Start 2006-10; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Total recovery at three months of onset, based on a global test analysis including NIHSS, mRS and Barthel Index | 3 months

SECONDARY OUTCOMES:
mRS at 3 months | 3 months
Barthel Index at 3 months | 3 months
Safety and tolerability | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Dávalos, MD, PhD, Study Chair — Hospital Universitari Germans Trias i Pujol, Badalona (Spain)
Locations (64):
- Germany (12):
  - Klinikum AltenburgerLand GmbH, Altenburg
  - Neurologie EVKB, Bielefeld
  - Neurologische Klinik Heinrich-Heine Universität, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Ernst-Moritz-Arndt-Universität Greifswald, Greifswald
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Neurologische Klinik Universitatsklinikum Heidelberg, Heidelberg
  - Klinikum Ingolstadt, Ingolstadt
  - Universitätsklinikum Leipzig, Leipzig
  - Johannes Wesling Klinikum Minden, Minden
  - Klinikum Großhadern der Universität München, München
  - Universitätsklinikum Münster, Münster
- Portugal (14):
  - Hospital de Sao Jose, Lisbon, Lisbon District
  - Hospital de Sao Joao, Porto, Porto District
  - Hospital Garcia de Orta, EPE, Almada
  - Hospital Garcia de Orta, Almada
  - Hospital Fernando Fonseca, Amadora - Sintra
  - Hospital Sao Marcos, Braga
  - Hospitais da Universidade Coimbra, Coimbra
  - Centro Hospitalar de Coimbra, Coimbra
  - Hospital de Santa Maria, Lisbon
  - Hospital de Santo Antonio, Porto
  - Hospital Sao Sebastiao, Santa Maria da Feira
  - Centro Hospitalar de Setúbal, EPE, Setúbal
  - Centro Hospitalar de Setúbal, Setúbal
  - Hospital Sao Pedro, Vila Real
- Spain (38):
  - Hospital General de Albacete, Albacete, Albacete
  - Hospital Son Dureta, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital de la Santa Creu I Sant Pau, Barcelona, Barcelona
  - Hospital Sagrat Cor, Barcelona, Barcelona
  - Hospital Vall d´Hebron, Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Mataro, Mataró, Barcelona
  - Consorci Hospitalari Parc Tauli, Sabadell, Barcelona
  - Hospital Moises Broggi, Sant Joan Despí, Barcelona
  - Hospital General Yague, Burgos, Burgos
  - Hospital San Pedro de Alcantara, Cáceres, Caceres
  - Hospital de Girona Dr. Josep Trueta, Girona, Girona
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital de Leon, León, Leon
  - Hospital Arnau de Vilanova, Lleida, Lleida
  - Complejo Hospitalario Xeral Calde, Lugo, Lugo
  - Hospital de La Princesa, Madrid, Madrid
  - Hospital Universitario Gregorio Marañon, Madrid, Madrid
  - Hospital Ramon y Cajal, Madrid, Madrid
  - Hospital Clinico San Carlos, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Central de Defensa (del Aire), Madrid, Madrid
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital Meixoeiro, Vigo, Pontevedra
  - Hospital Virgen Macarena, Seville, Sevilla
  - Hospital Universitario Virgen del Rocio, Seville, Sevilla
  - Hospital Universitario Nuestra Señora De Valme, Seville, Sevilla
  - Hospital Universitario La Fe, Valencia, Valencia
  - Hospital Clinico Universitario, Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario, Valladolid, Valladolid
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Marqués de Valdecilla, Santander
  - Hospital Clínico de Valladolid, Valladolid

REFERENCES:
- [Background] Bolland K, Whitehead J, Cobo E, Secades JJ. Evaluation of a sequential global test of improved recovery following stroke as applied to the ICTUS trial of citicoline. Pharm Stat. 2009 Apr-Jun;8(2):136-49. doi: 10.1002/pst.344. PMID 18637642
- [Result] Davalos A, Alvarez-Sabin J, Castillo J, Diez-Tejedor E, Ferro J, Martinez-Vila E, Serena J, Segura T, Cruz VT, Masjuan J, Cobo E, Secades JJ; International Citicoline Trial on acUte Stroke (ICTUS) trial investigators. Citicoline in the treatment of acute ischaemic stroke: an international, randomised, multicentre, placebo-controlled study (ICTUS trial). Lancet. 2012 Jul 28;380(9839):349-57. doi: 10.1016/S0140-6736(12)60813-7. Epub 2012 Jun 11. PMID 22691567